CLINICAL TRIAL: NCT06343441
Title: A Randomized Controlled, Double-blind Clinical Trial to Evaluate the Clinical Effectiveness of Two Methods of Taking Impressions for an Implant-supported Fixed Prostheses With One-piece Titanium Frameworks in Edentulous Jaws
Brief Title: Accuracy of Two Methods of Making Impressions for Complete-arch Implant Supported Fixed Prosthesis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Junyu Shi, Associate researcher, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SH9H-2024-T29-2
Record Dates: First submitted 2024-03-20; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Edentulous Jaw
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- digital impression (Experimental): intraoral scan
  Interventions: Device: intraoral scan
- conventional impression (Active Comparator): open tray
  Interventions: Device: open tray impression

INTERVENTIONS:
Device: intraoral scan — intraoral scanning of the edentulous arch and scan body
  Arms: digital impression
Device: open tray impression — conventional method of impression making with silicone rubber material
  Arms: conventional impression

SUMMARY:
To compare the accuracy of digital impression and conventional impression for complete-arch implant-supported fixed prosthesis

DETAILED DESCRIPTION:
The Intraoral scan is digital optical scan method, that has advantages such as being more comfortable, easy to transfer, and full digital workflow. Conventional impression using silicon rubber and gained stable accuracy of impression. This study aims to compare the accuracy of two methods.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old (including 18 and 70 years old);
* The patient's maxilla or mandible cannot be preserved due to missing teeth or remaining teeth proposed for implant-retained restoration;
* The patient's missing teeth area is available for placement of 4-6 implants;
* Completion of osseointegration of the patient's implants after implant surgery;
* The patient has at least 2 mm width of keratinized mucosa in the remaining alveolar ridge;
* The patient voluntarily participates in the trial and signs an informed consent form

Exclusion Criteria:

* The patient has a severe gag reflex;
* The patient has an intermaxillary distance of less than 20 mm in the posterior region;
* The distance between the two implants is less than 10 mm;
* Implants fitted with composite abutments with the abutment screw holes penetrating at an angle greater than 60 degrees to the alveolar ridge;
* Other patients judged by the investigator to be unsuitable for inclusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-03-31 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Grade of framework passive fit | during the deliver of the framework
  The passive fit of the titanium framework is measured with a scoring system. Five aspects are evaluated. whether to pry; Single Screw Probing misfit; All Screws; Probing misfit; Smooth during screwing; X-ray for misfit. For each aspect, 0/1 is scored. the total score is between 0 and 5.